CLINICAL TRIAL: NCT06675591
Title: Mortality and Neurologic Complications Associated With Rapid Versus Slow Correction of Hyponatremia
Brief Title: Mortality and Neurologic Outcomes in Rapid vs. Slow Hyponatremia Correction
Acronym: RASC-HypoNa
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: University of California, Irvine (Other); Hospital Privado de Comunidad de Mar del Plata (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, ANACLARA MURUJOSA, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 6756; 10042 (Other: PRIISA)
Record Dates: First submitted 2024-09-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Hyponatremia; Hospitalisation; Mortality; SEVERE HYPONATREMIA
Keywords: severe hyponatremia; sodium correction; Osmotic Demyelination Syndrome; rapid sodium correction; In-Hospital Mortality; cohort study
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rapid group correction: Patients whose serum sodium increased by ≥ 8 mEq/L within the first 24 hours.
  Interventions: Other: Rapid sodium correction
- Slow group correction: Patients whose serum sodium increased by < 8 mEq/L within the first 24 hours.
  Interventions: Other: Slow sodium correction

INTERVENTIONS:
Other: Rapid sodium correction — This study focuses on the exposure to different sodium correction rates in patients with severe hyponatremia (serum sodium ≤ 120 mEq/L) rather than an active intervention. The two key groups are defined by their rate of sodium correction during the first 24 hours of hospitalization:
  Rapid Sodium Correction: An increase in serum sodium of ≥ 8 mEq/L within 24 hours.
  Slow Sodium Correction: An increase in serum sodium of < 8 mEq/L within 24 hours.
  The primary objective is to assess the association between these exposure rates and clinical outcomes, including in-hospital mortality, 30-day mortality, and the incidence of osmotic demyelination syndrome (ODS). This study differs from others by using a large, retrospective cohort of patients treated in a real-world clinical setting, spanning 13 years (2010-2023), and applying robust statistical adjustments such as propensity score analysis to control for confounders.
  Groups: Rapid group correction
Other: Slow sodium correction — This study focuses on the exposure to different sodium correction rates in patients with severe hyponatremia (serum sodium ≤ 120 mEq/L) rather than an active intervention. The two key groups are defined by their rate of sodium correction during the first 24 hours of hospitalization:
  Rapid Sodium Correction: An increase in serum sodium of ≥ 8 mEq/L within 24 hours.
  Slow Sodium Correction: An increase in serum sodium of < 8 mEq/L within 24 hours.
  The primary objective is to assess the association between these exposure rates and clinical outcomes, including in-hospital mortality, 30-day mortality, and the incidence of osmotic demyelination syndrome (ODS). This study differs from others by using a large, retrospective cohort of patients treated in a real-world clinical setting, spanning 13 years (2010-2023), and applying robust statistical adjustments such as propensity score analysis to control for confounders.
  Groups: Slow group correction

SUMMARY:
This study examines the impact of different rates of sodium correction on the outcomes of patients with severe hyponatremia (serum sodium ≤ 120 mEq/L). Hyponatremia is a condition where blood sodium levels are dangerously low, and its treatment must be carefully managed to avoid complications. Standard guidelines recommend correcting sodium levels slowly to prevent a rare but serious neurological condition called osmotic demyelination syndrome (ODS). However, recent evidence suggests that a faster rate of sodium correction may reduce hospital stay length and mortality without increasing the risk of ODS.

This retrospective study, conducted from 2010 to 2023 at a hospital in Buenos Aires, Argentina. It compares the outcomes of patients who had their sodium levels corrected rapidly (≥ 8 mEq/L in 24 hours) to those who had slower corrections. The primary outcomes measured are mortality and the development of ODS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* First hospitalization at Hospital Italiano de Buenos Aires with a serum sodium (natremia) level ≤ 120 mEq/L at admission.

Exclusion Criteria:

* Absence of serum sodium values after the first 24 hours of hospitalization.
* Hospitalizations shorter than 24 hours.
* Patients with previous hospitalizations prior to the study period where admission serum sodium levels were ≤ 120 mEq/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older who were admitted to Hospital Italiano de Buenos Aires between 2010 and 2023 with severe hyponatremia, defined as a serum sodium (natremia) level of ≤ 120 mEq/L at the time of admission. The study focuses on patients experiencing their first hospitalization for this condition, with a hospital stay exceeding 24 hours to ensure sufficient follow-up for sodium correction. Patients with prior hospitalizations for severe hyponatremia or incomplete follow-up data were excluded to ensure accurate analysis of treatment outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 2037 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
In-Hospital Mortality | From hospital admission to discharge or death. To evalute in-Hospital mortality we will use logistic regression, not time to event analysis.
  In-Hospital Mortality refers to the occurrence of death from any cause during a patients hospital stay. In the context of this study, it specifically measures the rate at which patients with severe hyponatremia (serum sodium ≤ 120 mEq/L) die before being discharged from the hospital.

SECONDARY OUTCOMES:
30-Day Mortality | From the date of hospital admission up to 30 days. From hospital admission to discharge or death. To evalute 30-Day mortality we will use logistic regression, not time to event analysis.
  30-Day Mortality refers to the occurrence of death from any cause within 30 days following a patient's admission to the hospital. In this study, it measures the mortality rate of patients with severe hyponatremia (serum sodium ≤ 120 mEq/L) within 30 days after hospitalization, regardless of whether they were discharged or remained in the hospital.
Length of stay | From the date of hospital admission to the date of discharge
  Length of Stay (LOS) refers to the duration of a patient's hospitalization, measured from the date of admission to the date of discharge. In this study, it evaluates how long patients with severe hyponatremia (serum sodium ≤ 120 mEq/L) remain in the hospital and assesses whether the rate of sodium correction (rapid vs. slow) influences their hospital stay.
Incidence of Osmotic Demyelinitation Syndrome (ODS) | From the date of hospital admission through hospital discharge, up to 180 days.
  Incidence of Osmotic Demyelination Syndrome (ODS) refers to the number of new cases of ODS that occur in patients during or after the correction of severe hyponatremia (serum sodium ≤ 120 mEq/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoorn EJ, Halperin ML, Zietse R. Diagnostic approach to a patient with hyponatraemia: traditional versus physiology-based options. QJM. 2005 Jul;98(7):529-40. doi: 10.1093/qjmed/hci081. Epub 2005 Jun 13. PMID 15955797
- [Background] Whelan B, Bennett K, O'Riordan D, Silke B. Serum sodium as a risk factor for in-hospital mortality in acute unselected general medical patients. QJM. 2009 Mar;102(3):175-82. doi: 10.1093/qjmed/hcn165. Epub 2008 Dec 23. PMID 19106156
- [Background] Kovesdy CP, Lott EH, Lu JL, Malakauskas SM, Ma JZ, Molnar MZ, Kalantar-Zadeh K. Hyponatremia, hypernatremia, and mortality in patients with chronic kidney disease with and without congestive heart failure. Circulation. 2012 Feb 7;125(5):677-84. doi: 10.1161/CIRCULATIONAHA.111.065391. Epub 2012 Jan 5. PMID 22223429
- [Background] Mohan S, Gu S, Parikh A, Radhakrishnan J. Prevalence of hyponatremia and association with mortality: results from NHANES. Am J Med. 2013 Dec;126(12):1127-37.e1. doi: 10.1016/j.amjmed.2013.07.021. PMID 24262726
- [Background] Heuman DM, Abou-Assi SG, Habib A, Williams LM, Stravitz RT, Sanyal AJ, Fisher RA, Mihas AA. Persistent ascites and low serum sodium identify patients with cirrhosis and low MELD scores who are at high risk for early death. Hepatology. 2004 Oct;40(4):802-10. doi: 10.1002/hep.20405. PMID 15382176
- [Background] Abebe TB, Gebreyohannes EA, Tefera YG, Bhagavathula AS, Erku DA, Belachew SA, Gebresillassie BM, Abegaz TM. The prognosis of heart failure patients: Does sodium level play a significant role? PLoS One. 2018 Nov 8;13(11):e0207242. doi: 10.1371/journal.pone.0207242. eCollection 2018. PMID 30408132
- [Background] Xiao M, Wang X, Wang H, Du F, Yao Y, Wang X, Wang J, Yang J, Xiong W, Wang Q, Ren X, Zhu T. Risk factors for hyponatremia in acute exacerbation chronic obstructive pulmonary disease (AECOPD): a multicenter cross-sectional study. BMC Pulm Med. 2023 Jan 28;23(1):39. doi: 10.1186/s12890-023-02328-4. PMID 36709254
- [Background] Seethapathy H, Zhao S, Ouyang T, Passos C, Sarang A, Cheung PW, Waikar SS, Steele DJR, Kalim S, Allegretti AS, Ayus JC, Nigwekar SU. Severe Hyponatremia Correction, Mortality, and Central Pontine Myelinolysis. NEJM Evid. 2023 Oct;2(10):EVIDoa2300107. doi: 10.1056/EVIDoa2300107. Epub 2023 Sep 26. PMID 38320180
- [Background] Kinoshita T, Mlodzinski E, Xiao Q, Sherak R, Raines NH, Celi LA. Effects of correction rate for severe hyponatremia in the intensive care unit on patient outcomes. J Crit Care. 2023 Oct;77:154325. doi: 10.1016/j.jcrc.2023.154325. Epub 2023 May 13. PMID 37187000